CLINICAL TRIAL: NCT05130632
Title: Combustion of Plastic Waste and Human Health Effects in Guatemala
Brief Title: Plastic Waste and Human Health Effects in Guatemala
Acronym: Ecolectivos
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Universidad del Valle, Guatemala (Other); University of California, San Francisco (Other); University of Georgia (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Lisa M. Thompson, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002412; R01ES032009 (NIH); 1F31ES036126 (NIH); 1P2CES033430-01 (NIH)
Record Dates: First submitted 2021-10-20; First posted 2021-11-23 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Environmental Exposure
Keywords: Plastic Burning Practice; Plastic Waste Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The community working group (Experimental): Female participants over the age of 15 randomized to the intervention group will participate in working group sessions over 12 weeks' time that addresses plastic waste and introduce strategies to reduce use, recycle, and repurpose plastic. Community members of participants in the intervention group will also be invited to participate in the working groups.
  Interventions: Behavioral: The community working group
- Control Group. (No Intervention): Participants in control villages will receive small trees for reforestation during the intervention activities in the intervention group.

INTERVENTIONS:
Behavioral: The community working group — The intervention consists of educational working group (WG) sessions over 12 weeks. Eight core modules discussing essential elements (such as main problems of solid waste management, health effects of exposure to burning plastic, sustainable alternatives to plastic litter) and four periphery modules to help identify community-driven interventions to reduce plastic burning in household fires, consume less plastic, recycle, and repurpose plastic, will be held.
  Participants will prioritize one task that can be attained in the next 9 months, with the guidance of community workers (promotoras), such as:
  * engaging in a community clean-up
  * starting an organic compost pile free of plastic waste
  * training on community recycling, focusing on plastics recycling
  * making organic soaps, to use for personal grooming or washing clothes, eliminating plastic packaging
  * creating materials out of plastic, like bottle planters
  Other Names: Intervention Group
  Arms: The community working group

SUMMARY:
Ecolectivos is a type-1 hybrid-effectiveness-implementation study that uses a village-level cluster randomized controlled trial design. The goal of this study in rural Guatemala is to assess intervention strategies to reduce plastic burning in 8 intervention villages compared to 8 control villages. The intervention group participants will participate in 12 weekly behavioral working group sessions; the control group will not receive any specific activities. Two hundred women of reproductive age and other community members from these villages will be enrolled in each group. The follow-up period is 12 months. Data will be collected via interviews, focus groups, air pollution sampling, plastic waste collection, urinary biomarker assessments, and ambient air sampling. Program evaluation and results dissemination will occur in the last year of the project.

DETAILED DESCRIPTION:
Household air pollution from solid fuel combustion (e.g., wood) is a major environmental risk factor in low- and middle-income countries, accounting for an estimated 2.6 million deaths annually (World Health Organization, 2018). The contribution of plastic waste incineration in household fires has not been quantified. This is problematic for countries like Guatemala, where 71% of households burn waste as a primary means of disposal (Government of the Republic of Guatemala 2019). Plastic waste incineration is a critical, but understudied, public health and environmental hazard, as communities are inundated with cheap plastic without the means of safely disposing of plastic waste.

This study aims to conduct a type 1 hybrid-effectiveness-implementation study that uses a village-level cluster-randomized controlled trial design to evaluate the uptake and sustainability of intervention strategies to reduce the use, recycling, and repurposing of plastic that will lead to reductions in household-level plastic burning in selected villages in rural Guatemala. The 200 intervention group participants and other interested community members will participate in 12 weekly behavioral working group sessions. Each intervention community will commit to alternatives to burning plastic and drive initiatives they can achieve over the next 9 months. The 200 control group participants will not receive any specific activities until year 5, when dissemination of results will include control villages. Primary endpoints include personal exposure to air pollution, including particulate matter, black carbon, and other compounds produced while burning solid fuels and plastic waste. Secondary endpoints are assessed using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) implementation science framework.

ELIGIBILITY:
Inclusion Criteria:

For attendees at community working groups:

* There are no inclusion or exclusion criteria as the whole community will be invited

For questionnaires administered to workshop attendees:

* Over the age of 15

For the collection of urine and personal air pollution samples:

* Women of reproductive age (15 - <44 years, verified by official document)
* Willingness to attend 12-week working groups
* Willingness to participate in biomonitoring
* Willingness to wear a silicone wristband for 1 week at baseline and 4-5 months
* Household uses biomass as the primary fuel for cooking
* Reports daily participation in household cooking
* Reports that plastic is burned in household fires at least once a week (in the cooking stove or outdoors)
* Plans to live in the household for the next 12 months

For promotoras:

* Over the age of 18
* Ability to read and write
* Women who participate in biomonitoring in the intervention group
* Willingness to make monthly household visits to study participants
* Willingness to make weekly calls to study participants
* Willingness to encourage participation in the activity selected by the village
* Willingness to communicate weekly with the research team
* Willingness to support community meetings to scale up the intervention in intervention and control villages

Exclusion Criteria:

* Inability to consent
* Cognitively impaired or individuals with impaired decision-making capacity
* Pregnant women. However, women who become pregnant during the study may continue to participate.
* Women who report using tobacco products

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in PM2.5 exposure | Baseline, 4-5 months, and up to 13 months
  Air pollution exposure will be assessed using repeated 24-hour measurements. This study will compare differences in personal PM2.5 exposure among women participating in the two study arms.
Change in black carbon (BC) exposure | Baseline, 4-5 months, and up to 13 months
  Air pollution exposure will be assessed using repeated 24-hour measurements. This study will compare differences in personal BC exposure among women participating in the two study arms.
Change in urinary bisphenols | Baseline, 4-5 months, and up to 13 months
  To assess urinary biomarkers of exposure to plastic combustion, this study will compare differences in bisphenol concentrations among women participating in the two study arms.
Change in urinary phthalates | Baseline, 4-5 months, and up to 13 months
  To assess urinary biomarkers of exposure to plastic combustion, this study will compare differences in phthalate concentrations among women participating in the two study arms.
Change in urinary polycyclic aromatic hydrocarbons (PAHs) | Baseline, 4-5 months, and up to 13 months
  To assess urinary biomarkers of exposure to combustion by-products, including plastic, this study will compare differences in PAH concentrations among women participating in the two study arms.
Change in urinary volatile organic compounds (VOCs) | Baseline, 4-5 months, and up to 13 months
  To assess urinary biomarkers of exposure to combustion by-products, including plastic, this study will compare differences in VOC concentrations among women participating in the two study arms.

SECONDARY OUTCOMES:
Reach of intervention using the RE-AIM implementation science framework | 4-5 months and up to 13 months
  Using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) implementation science framework, assess the reach of the intervention in the intervention arm, as measured by: 1) the number and proportion of total invited participants who attend working groups; 2) the number and proportion of participants' household members who engage in working group activities; and 3) the number of intervention village members who engage in working group activities.
Effectiveness of intervention using the RE-AIM implementation science framework | 4-5 months and up to 13 months
  Using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) implementation science framework, assess the effectiveness of the intervention by measuring the number of intervention group participants who report behavior changes. These changes are categorized as "high" or "low" behaviors based on factors such as working group attendance, engagement in activities, and reported reductions in plastic burning.
Enablers and barriers to the adoption of the intervention using the RE-AIM implementation science framework | 13 months
  Using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM implementation science framework, assess the enablers and barriers to the adoption of the intervention using qualitative data collected from focus groups and interviews with participants and environmental promotoras. This will help identify the factors influencing the uptake of the intervention at the village level. There are no units of measure.
Adoption of the intervention by direct observation using the RE-AIM implementation science framework | 13 months
  Using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) implementation science framework, assess the adoption of the intervention through direct observations of intervention activities, using qualitative data analysis to evaluate the extent of implementation at the community level. There are no units of measure.
Maintenance of the intervention using the RE-AIM implementation science framework | After 13 months
  Using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) implementation science framework, assess the maintenance (sustainment of intervention strategies) at the participant, household, and village level, as measured by: 1) number and proportion of participants who report no longer burning plastic in household fires (a measure of de-adoption); 2) number and proportion of households who continue their involvement in intervention activities at the village level after the working groups are completed; and 3) number of community members and organizations who have independently maintained, or established, similar intervention activities in the communities after the working groups are completed in the intervention arm.

OTHER OUTCOMES:
Change in Health-related Quality of Life (HRQOL) Score | Baseline, 4-5 months, and up to 13 months
  Using the HRQOL instrument, compare differences in quality of life among women participating in the two study arms. The HRQOL consists of 4 questions measuring: a) overall general health (5 items- excellent, very good, good, fair, or poor; used independently, ordinal outcome); b) number of days physical health was not good in the last 30 days; c) number of days mental health was not good in the last 30 days (b and c are summed together, not to exceed 30 days, continuous outcome); and d) number of days poor physical or mental health limited daily activities in the last 30 days (used independently, continuous outcome). Higher scores typically represent poorer health and quality of life, with individuals reporting more health-related problems and worse functioning in daily activities, mental well-being, and social interactions. Lower scores suggest better health status, with individuals reporting fewer limitations or challenges in their physical, emotional, or social well-being.
Change in Household Decision Making | Baseline, 4-5 months, and up to 13 months
  Using a 7-part instrument, compare differences in household decision-making (e.g., spending earned money, major and minor purchases, job decisions, cooking foods, visiting others) among women participating in the two study arms. The responses are coded on a 4-point scale (respondent's sole decision; husband's decision; joint decision between respondent and husband; other family member makes decision). Scores range from 7 to 28; the lower the score, the greater the woman's agency to make household decisions.
Change in New General Self-Efficacy Scale (NGSE) Score | Baseline, 4-5 months, and up to 13 months
  Using the New General Self-Efficacy Scale (NGSE), an 8-part instrument, compare differences in self-efficacy (e.g., problem-solving, goal setting, confidence, resourcefulness) among women participating in the two study arms. Each item is rated on a 5-point scale (strongly disagree; disagree; neither agree nor disagree; agree; strongly agree). NGSE scores range from 5 to 40; the higher the score, the greater the individual's generalized self-efficacy belief.
Change in Short Social Capital Assessment Tool (SASCAT) Score | Baseline, 4-5 months and up to 13 months
  Using the 12-part Short Social Capital Assessment Tool, compare differences in group membership, citizenship, and cognitive social capital (trust) among women participating in the two study arms. Responses are Yes/No, and scoring ranges from 0-37. The responses are summed to calculate a total social capital score, with higher scores indicating higher levels of social capital, signifying more support, trust, and participation in community networks.
Change in Community Mobilization Scale Score | Baseline, 4-5 months and up to 13 months
  Using the Community Mobilization Scale, compare differences in the Critical Consciousness sub-scale (modified 9-item instrument) and the Collective Action sub-scale (modified 2-item instrument) among women participating in the two study arms. The Critical Consciousness sub-scale score is measured using a 3-point Likert scale (agree, somewhat agree, disagree; scores ranging from 9-27, measured continuously). The Collective Action sub-scale asks about the number of times the participant and community have worked on community problems in the last 3 months and is measured continuously. For both scales, higher scores indicate higher levels of mobilization.
Change in the quantification of emissions estimates of air pollutants from plastic incineration. | Baseline, 4-5 months and up to 13 months
  Using filter-based antimony (Sb) and 1,3,5-Triphenylbenzene (TPB) as tracers of plastic burning and collecting household plastic waste, apportion PM2.5 and quantify emissions estimates of air pollutants from plastic incineration and assess effects of potential emissions reduction on air quality with a chemical transport model.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Thompson, PhD, RN, FNP, Principal Investigator — Emory University - Nell Hodgson Woodruff School of Nursing; Eri Saikawa, PhD, Principal Investigator — Emory College of Arts and Sciences: Environmental Sciences
Locations (2):
- Guatemala (2):
  - Universidad del Valle de Guatemala, Guatemala City
  - Project Office, Jalapa, Jalapa

IPD SHARING:
Plan to Share IPD: Yes
Plan to share the following information: Exposure data, laboratory data, questionnaire related to the outcome and intervention, and standard of operating procedures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after the study ends or when submitting publication (at editor's or funder's request)
Access Criteria: The research team will create a data request form where they will outline procedures for accessing de-identified data which will include the name and affiliation of researchers, outcomes, and variables being requested with an approved statistical analysis plan.

REFERENCES:
- [Derived] Thompson LM, Lovvorn AE, Raheel H, Hengstermann-Artiga M, Lopez MR, Ramirez A, Barr DB, Higgins M, McCracken JP, Saikawa E, Handley MA. A village-level cluster randomized controlled implementation trial to measure the effectiveness of a behavioral intervention aiming to reduce women's exposures to household plastic waste burning in rural Guatemala: study protocol for the Ecolectivos trial. Trials. 2025 Dec 13. doi: 10.1186/s13063-025-09338-z. Online ahead of print. PMID 41390662

DOCUMENTS (1):
  • Informed Consent Form (2024-04-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT05130632/ICF_000.pdf